CLINICAL TRIAL: NCT02787161
Title: Impact of HemoDiaFIltration on Physical Activity and Self-reported Outcomes: a Randomized Controlled Trial (HD-FIT Trial)
Brief Title: Impact of HemoDiaFIltration on Physical Activity and Self- Reported Outcomes
Acronym: HDFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontifícia Universidade Católica do Paraná (Other)
Collaborators: Fresenius AG (Industry)
Responsible Party: Principal Investigator, Roberto Pecoits-Filho, MD, PhD, FASN, FACP, Pontifícia Universidade Católica do Paraná
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUCPR02
Record Dates: First submitted 2016-04-20; First posted 2016-06-01 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Hemodialysis; Hemodiafiltration; Renal Replacement Therapy; Physical Activity; Accelerometer
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity | interventions — Hemodiafiltration; Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemodialysis (Active Comparator): Patients who are treated with high flux hemodialysis will continue the same treatment with high flux hemodialysis.
  Interventions: Device: Hemodialysis
- Hemodiafiltration (Experimental): Patients who are treated with high flux hemodialysis will be switched to hemodiafiltration for 6 months.
  Interventions: Device: Hemodiafiltration

INTERVENTIONS:
Device: Hemodiafiltration — High volume online HDF
  Other Names: High volume online HDF
  Arms: Hemodiafiltration
Device: Hemodialysis — High-flux HD
  Other Names: High-flux HD
  Arms: Hemodialysis

SUMMARY:
This is a randomized controlled clinical trial that will analyze the impact of high volume online HDF in comparison to high-flux HD on measured physical activity.

DETAILED DESCRIPTION:
HD-FIT is a randomized controlled clinical trial that will analyze the impact of high volume online HDF in comparison to high-flux HD on measured physical activity (number of steps measured in the dialysis day) as a primary endpoint. The analysis of additional accelerometer data, HRQOL and time to recover from a dialysis session will be used as other outcomes. The study will also capture safety data, based on intradialytic events, hospitalization and mortality. Biochemical (according to the local requirements) and drug prescription data will be monitored for pharma-economic analysis. Serum samples will be collected for future analysis of additional biomarkers.

In summary, patients will go through a 4 week run in period on high flux HD. After this, patients will be randomized to the intervention of high volume online HDF for 6 months, or will continue on high flux HD; both groups will be observed for a 12 month follow up period. Patients will be evaluated for physical activity, HRQOL, laboratories and other measures at the baseline, 3 month, and 6 month time points. Evaluation will be repeated in 3 and 6-months. HRQOL, laboratories, and other outcomes will be tracked over the post-interventional follow up period that lasts 12 months after randomization.

Data will be analyzed according to an intention-to-treat principle (i.e., according to assigned instead of received treatment). With an enrollment target of 110 participants in each arm (considering a drop out of 20%) we estimate the 86 patients will complete the follow up in each arm, what will provide the trial a 90% power to detect a 20% effect with respect to the primary outcome (predefined as a 20% increase in average total steps at the dialysis day in the HDF group compared to the HD group). Because of the nature of the intervention, it will not possible to blind the patients, the local study nurses, or the investigators for the treatment assignment.

Fourteen dialysis centers will be invited to participate. Each participating center will receive two 5008S machines and Cordiax dialyzers to be used in the study of 10 patients in each center. Additional patients can be randomized per center with approval of the steering committee. Centralized randomization will based on a 1:1 protocol, stratified by participating center.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated three times per week with HD for at least 3 months and up to 24 months;
* Clinically stable according to the evaluation of the investigator;
* Kt/V of > 1.2;
* Patients with an arteriovenous fistula/graft and permanent catheters with adequate flow.

Exclusion Criteria:

* Age below 18 years;
* Life expectancy less than 3 months because of nonrenal disease;
* Participation in another clinical intervention trial;
* Severe non-compliance regarding frequency and duration of dialysis treatment;
* Patients with severe limitation to mobility (amputated, neurologic and muscular disorders) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
The difference in the change in step counts per 24 hours on dialysis days from baseline to the 6-month follow up in patients treated with high volume online HDF versus high-flux HD | Baseline, 3 months and 6 months
  To capture activity in the study, we will use the Actigraph ™ device to measure acceleration and count steps during 7 days at baseline, 3 and 6 months evaluations, according to a previously described protocol for dialysis patients. A 4s step filter is an intrinsic property of the Actigraph ™ that screens out erroneous steps that might result as from shuffling, standing up, sitting up, sitting down, and vibrations from a moving vehicle. The Actigraph ™ is lightweight (19g), clips at the waist, and provides feedback with on-instrument digital display of step counts. It interfaces with the internet via bluetooth, allowing upload of date and time stamped step counts.
The difference in the change in minutes of moderate-to-vigorous physical activity (MVPA) per 24 hours on dialysis days from baseline to the 6-month follow up in patients treated with high volume online HDF versus high-flux HD | Baseline, 3 months and 6 months

SECONDARY OUTCOMES:
The difference in the change in self-reported dialysis recovery time from baseline to the 6-month follow up in patients treated with high volume online HDF versus high-flux HD | Baseline, 3 months and 6 months
  Dialysis recovery time will be assessed at baseline and at 3 and 6 months of follow-up in both arms. The dialysis recovery time survey asks the question, " How long does it take to recover from a dialysis session?" . This test has been validated in HD studies, and it is interpreted easily, is easy to respond to, shows stability over time by test-retest, shows both convergent and divergent validity, and is sensitive to change.
The difference in the change in SF-36 scores from baseline to the 6-month follow up in patients treated with high volume online HDF versus high-flux HD | Baseline, 3 months and 6 months
  HRQOL will be assessed at baseline and at 3 and 6 months of follow- up with the Kidney Disease Quality of Life - Short Form (KDQOL-SF), adapted and validated to Brazilian Portuguese. This questionnaire covers different domains to face the multidimensional nature of HRQOL. The eight domains of the SF-36 can be summarized in two summary scores, one for physical functioning (the physical composite score [ PCS]) and one for mental functioning (the mental composite score [MCS]). Questionnaires will be applied at the baseline, and 3 and 6 months in both arms. Analysis will include PCS and MCS.
Pharmacoeconomy (drug use, hospitalization) | Baseline, 3 months and 6 months
  Income, social status, prescription of drugs, hospitalization
Intradialytic events | Baseline, 3 months and 6 months
  Events
Mortality | Baseline, 3 months and 6 months
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Flávio Pecoits-Filho, PI, Study Chair — PUC-PR
Locations (13):
- Brazil (13):
  - Instituto Médico Nefrológico, Belo Horizonte, Minas Gerais
  - Nefron Contagem, Contagem, Minas Gerais
  - Irmandade da Santa Casa de Misericórdia de Curitiba, Curitiba, Paraná
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundação Pro Rim, Joinville, Santa Catarina
  - Instituto de Nefrologia de Taubaté, Taubaté, São Paulo
  - Clínica de Diálise Ingá, Rio de Janeiro
  - Clínica de Doenças Renais - São Lourenço, Rio de Janeiro
  - Clínica de Doenças Renais - Un. Botafogo, Rio de Janeiro
  - CETENE, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital do Rim e Universidade Federal de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lima JD, Guedes M, Rodrigues SD, Florido ACS, Moreno-Amaral AN, Barra AB, Canziani ME, Cuvello-Neto A, Poli-de-Figueiredo CE, Pecoits-Filho R, Nakao LS. High-volume hemodiafiltration decreases the pre-dialysis concentrations of indoxyl sulfate and p-cresyl sulfate compared to hemodialysis: a post-hoc analysis from the HDFit randomized controlled trial. J Nephrol. 2022 Jun;35(5):1449-1456. doi: 10.1007/s40620-022-01283-3. Epub 2022 Mar 3. PMID 35239175
- [Derived] Guedes M, Dambiski AC, Canhada S, Barra ABL, Poli-de-Figueiredo CE, Cuvello Neto AL, Canziani MEF, Strogoff-de-Matos JP, Raimann JG, Larkin J, Canaud B, Pecoits-Filho R; HDFIT Study Investigators. Achieving high convective volume in hemodiafiltration: Lessons learned after successful implementation in the HDFit trial. Hemodial Int. 2021 Jan;25(1):50-59. doi: 10.1111/hdi.12891. Epub 2020 Oct 15. PMID 33058473
- [Derived] Larkin JW, Han M, Han H, Guedes MH, Goncalves PB, Poli-de-Figueiredo CE, Cuvello-Neto AL, Barra ABL, de Moraes TP, Usvyat LA, Kotanko P, Canziani MEF, Raimann JG, Pecoits-Filho R; HDFIT Study Investigators. Impact of hemodialysis and post-dialysis period on granular activity levels. BMC Nephrol. 2020 May 25;21(1):197. doi: 10.1186/s12882-020-01853-2. PMID 32450793
- [Derived] Pecoits-Filho R, Larkin JW, Poli-de-Figueiredo CE, Cuvello Neto AL, Barra AB, Canhada S, de Campos LG, Woehl J, Goncalves PB, Han H, de Moraes TP, Raimann JG, Canziani MEF; HDFIT Study Investigators. Design and methodology of the impact of HemoDiaFIlTration on physical activity and self-reported outcomes: a randomized controlled trial (HDFIT trial) in Brazil. BMC Nephrol. 2019 Mar 20;20(1):98. doi: 10.1186/s12882-019-1247-8. PMID 30894141